CLINICAL TRIAL: NCT05121402
Title: A Phase 2 Multicenter, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of TLL018 for Induction Therapy in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Safety and Efficacy Study of TLL018 in the Treatment of Ulcerative Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decisions made by senior management of the company
Sponsor: TLL Pharmaceutical, LLC (Industry)
Responsible Party: Sponsor
Organization: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLL018-202
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose TLL018,BID (Experimental): Drug: TLL018 all subjects will receive TLL018 for 8 weeks
  Interventions: Drug: TLL018
- Middle dose TLL018,BID (Experimental): Drug: TLL018 all subjects will receive TLL018 for 8 weeks
  Interventions: Drug: TLL018
- High dose TLL018,BID (Experimental): Drug: TLL018 all subjects will receive TLL018 for 8 weeks
  Interventions: Drug: TLL018
- Placebo (Placebo Comparator): Placebo twice daily for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TLL018 — a TYK2/JAK1 inhibitor
  Arms: High dose TLL018,BID; Low dose TLL018,BID; Middle dose TLL018,BID
Other: Placebo — a TLL018 Placebo
  Arms: Placebo

SUMMARY:
A study to investigate the safety and efficacy of TLL018 compared with placebo in subjects with moderate to severe ulcerative colitis.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, randomized, double-blind, parallel dose groups, placebo-controlled dose ranging study to evaluate the safety and efficacy of 3 doses of TLL018 as an induction therapy in subjects with moderate to severe UC.

Eligible subjects will be randomized to receive one of the following treatments: TLL018 low dose, TLL018 middle dose, TLL018 high dose, or placebo. All subjects may remain on a stable dose of conventional therapy used prior to enrollment. Subjects will be assessed for safety, tolerability, and response to treatment. Samples for pharmacokinetics (PK) and pharmacodynamics (PD) biomarker analyses will be collected throughout the study according to the Schedule of Assessments (SoA) for potential correlation to clinical outcomes.

Further participation may continue beyond the initial 8 weeks for another 5-week Extension Period of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 and ≤ 75 years of age at baseline.
* Capable of giving informed consent and complying with study procedures.
* Normal renal function or mild renal impairment as determined by the Investigator following review of clinical laboratory test results.
* Laboratory and medical history parameters within the protocol-defined ranges.
* Diagnosis of UC for 90 days or greater prior to baseline, confirmed by colonoscopy during the screening period, with exclusion of current infection, colonic dysplasia, and/or malignancy. Appropriate documentation of biopsy results consistent with the diagnosis of UC, in the assessment of the Investigator, must be available.
* Active UC with a full Mayo score of 6 to 12 points and endoscopic subscore of 2 or higher confirmed by central reader.
* Subject must have received COVID-19 vaccine >2 months before first dose of study drug.

Exclusion Criteria:

* Pregnant or nursing women.
* Clinically significant history of cardiovascular, hematologic, renal, hepatic, bronchopulmonary, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator.
* Current and/or recent history of a clinically significant infection.
* Any history of malignancies, except for non-melanoma skin cancers (unless it is metastatic).
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
* Any condition or finding that in the Investigator's opinion would put the subjects or study conduct at risk if the subjects were to participate in the study.
* Current diagnosis of Crohn's disease (CD) or diagnosis of indeterminate colitis (IC).
* Current diagnosis of fulminant colitis and/or toxic megacolon, or active Clostridium difficile colitis.
* Subject with disease limited to the rectum (ulcerative proctitis) during the screening endoscopy.
* Subject with previous exposure to JAK inhibitor (eg, tofacitinib, baricitinib, filgotinib, upadacitinib).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who achieved clinical remission per adapted Mayo score at Week 8 | Baseline to Week 8
Number of treatment-emergent adverse events (TEAEs) | Up to 8 weeks
  TEAE defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Incidence of Adverse Events (AEs) and Adverse Events of Special Interest (AESIs) | Up to 8 weeks
Number of Participants With Clinically Significant Changes in clinical laboratory data | Up to 8 weeks
  Laboratory investigation included hematology, biochemistry, urinalysis and coagulation. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in laboratory parameters were reported.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Up to 8 weeks
  Vital signs included body temperature, systolic and diastolic blood pressure, pulse rate, respiratory rate, weight and height. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in vital signs were reported.
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings | Up to 8 weeks
  Clinically significant ECG criteria included QT interval corrected using the Fridericia's formula (QTCF) value 450 msec and 30<=change<60.

SECONDARY OUTCOMES:
Percentage of subjects with endoscopic improvement at Week 8 | Week 8
Percentage of subjects with endoscopic remission at Week 8 | Week 8
Percentage of subjects achieving clinical response per adapted Mayo score at Week 8 | Week 8
Percentage of subjects achieving clinical response per partial adapted Mayo score at Week 2 | Week 2
Percentage of subjects who achieved histologic-endoscopic mucosal improvement (as defined by endoscopic subscore and Geboes score) at Week 8 | Week 8
Percentage of subjects with mucosal healing (as defined by the endoscopic and histologic variables) at Week 8 | Week 8
Percentage of subjects who achieved histologic improvement (as defined by Geboes score) at Week 8 | Week 8
Percentage of subjects who reported no bowel urgency (as monitored electronically via a handheld device) at Week 8 | Week 8
Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Score | Baseline to Week 8
  The IBDQ is used to measure disease specific quality of life on a 32 Likert-scaled items questionnaire. The IBDQ scale contains 4 component subscales: bowel symptoms, systemic symptoms, emotional function and social function with scores ranging from 10 to 70, 5 to 35, 12 to 84 and 5 to 35 respectively and the total score ranges from 32 to 224. Higher scores indicate better health related quality of life.
Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Questionnaire Score | Baseline to Week 8
  The FACIT system is a collection of quality of life (QOL) questionnaires targeted to the management of cancer and other chronic illnesses.
Time to improvement as measured by rectal bleeding via handheld device | Baseline to Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Research of San Antonio (GERSA), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided